CLINICAL TRIAL: NCT03265691
Title: Effectiveness of Early Intervention in the Diagnosis and Treatment of Hyponatremia in the Prevention of Hospitalized Patients Falls
Brief Title: Hyponatremia in the Prevention of Hospitalized Patients Falls
Acronym: PRECAHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mª del Carmen Lobo Rodríguez (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor-Investigator, Mª del Carmen Lobo Rodríguez, Msc Nurse Research, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: V01_Enf
Record Dates: First submitted 2016-05-10; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Hyponatremia; Accidental Falls
Keywords: Accidental Falls; Hyponatremia; Elderly; Risk factors; Nurse
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early hyponatremia diagnosis and treatment (Experimental): The early diagnosis of hiponatremia is not a stándar procedure. In the experimental arm, hyponatremia will be diagnosed and treated early.
  Interventions: Other: Early detection and treatment of hyponatremia; Other: No Intervention (SOC)
- No intervention (No Intervention): Usual pattern of work will be performed in all patients who enter in Hospital. Duration: 6 months.

INTERVENTIONS:
Other: Early detection and treatment of hyponatremia — In the experimental group, hyponatremia will be diagnosed and treated early. Therefore, the researchers will review the patients' sodium levels at admission and throughout their stay.
  Arms: Early hyponatremia diagnosis and treatment
Other: No Intervention (SOC) — Usual pattern of work will be performed in all patients who enter in Hospital.
  Arms: Early hyponatremia diagnosis and treatment

SUMMARY:
Cross ecological quasi-experimental study to assess effectiveness of early intervention in the diagnosis and treatment of hyponatremia in the prevention of hospitalized patients´ falls.

DETAILED DESCRIPTION:
Effectiveness of early intervention in the diagnosis and treatment of hyponatremia in the prevention of hospitalized patients´ falls.

Aims:

1. To assess the effectiveness of corrective activity of hyponatremia in falls reducing incidence.
2. To assess the cost-effectiveness ratio of the two proposed strategies: conventional treatment versus early intervention.

Cross ecological quasi-experimental study. The project will take place in Gregorio Marañón Hospital (Madrid, Spain) in the following inpatient adult Units: Neurology, Rehabilitation 1, Geriatrics, Internal Medicine (Group A), Cardiology, Rehabilitation 2, Gastroenterology, Neurosurgery and Oncology (Group B).

The estimated sample size for a confidence level of 95% (α = 0.05) and power of 90% (β = 0.010), taking into account a decrease in the incidence of falls of 20% restocking losses, is 124 patients per group (ie, the 124 patients receiving regular performance ** and 124 patients receiving the experimental intervention *, if necessary, by participant Unit).

Data collection: In each of the study participants Units both interventions will be held. First the participants Units have been randomized in two groups (Group A: Neurology, Rehabilitation 1, Geriatrics, Internal Medicine; Group B: Cardiology, Rehabilitation 2, Gastroenterology, Neurosurgery and Oncology). All patients hospitalized in these Units will be potentially included. First of all, collaborators will give them an informed consent to ask for their participation.

The interventions are:

* Experimental intervention: early diagnosis, treatment of hyponatremia until resolution and valuation according to the Dynamic Gait Index test. Duration: 6 months
* Habitual action: the usual pattern of work will be performed in all patients who enter. Duration: 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Admitted to a participating study unit
* Wish to participate in the study and signature of informed consent.

Exclusion Criteria:

* Transfer of the patient to a unit not included in the study
* Deterioration of the patient's condition to severe or extremely painful

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of treatment of hyponatremia in reducing the incidence of falls. | 1 year
  The effectiveness will be measured in terms of less incidence of falls

SECONDARY OUTCOMES:
To evaluate the cost-effectiveness of the 2 strategies proposed: conventional treatment vs early intervention. | 1 year
  The cost-effectiveness will be indirectly measured using Average cost per inpatient day

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Lobo-Rodriguez, pHd, Principal Investigator — carmen.lobo@salud.madrid.org
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No